CLINICAL TRIAL: NCT03720912
Title: Effect of Behavioral Family Therapy on Glycemic Control in Children With Type One Diabetes
Brief Title: Behavioral Family Therapy and Type One Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of Nevada, Reno (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1303325
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be masked to the participant's assignment. Others (participant, care provider, investigator) cannot be masked to assignment because one group will be receiving the behavioral health intervention and the other will not be receiving anything additional.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Family Education Modules (Experimental): Patients will receive online family education modules.
  Interventions: Behavioral: Online Learning Modules
- Control (No Intervention): Patients will not receive any intervention.

INTERVENTIONS:
Behavioral: Online Learning Modules — The modules will include information about common family management skills: social support, problem solving, communication, and supportive behavior change strategies.
  Arms: Online Family Education Modules

SUMMARY:
Behavioral family therapy, specifically focused on insuring support for the primary caregiver of a child with type one diabetes mellitus and healthy family dynamics, may improve the child's glycemic control as measured by hemoglobin A1c level (HbA1c).

DETAILED DESCRIPTION:
The success or failure of type 1 diabetes mellitus (T1D) management in children depends not only on access to care, diabetes technologies and diabetes education, but also on the abilities of the patient and his/her family to carry out complex demands. Recent data show that family dynamics play a critical role in determining glycemic control in pediatric patients with T1D. The investigators prior work (Loomba-Albrecht and Glaser, unpublished data) suggests that the strongest determinants of glycemic control are factors related to the primary caregiver's involvement in supportive relationships with others, either a spouse or other family members. This provides a potential therapeutic target to improve outcomes for children with T1D.

ELIGIBILITY:
Inclusion Criteria:

* age 2 to 17 years
* newly diagnosed (within the past 12 weeks) with T1D
* seeking care at UC Davis

Exclusion Criteria:

- Families will be excluded if the child has severe underlying psychiatric, behavioral or medical conditions which could independently affect parental marital stress

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c Level | 6, 12, 18, and 24 months
  The main outcome variable will be the change in glycemic control measured as the mean HbA1c level over the two years following study enrollment.

SECONDARY OUTCOMES:
Behavioral Affect Rating | At enrollment and approximately 3 months after enrollment
  22 item assessment of the level of hostility and warmth/supportiveness that each parent has received from his or her partner over the prior month-married parents will complete; Scale range is 1 (always)-7 (never); sclae is divided into two parts, hostility and warmth/support (higher values indicate higher hostility or higher warmth/support)
Child Perception of Interparental Conflict (CPIC) | At enrollment and approximately 3 months after enrollment
  Child's assessment of conflict between parents (completed by children ages 6-18 years of married parents); scale range is 1 (best)-5 (worst), Questions 1 and 4 are reverse scored
Family Assessment Device-General Functioning Subscale | At enrollment and approximately 3 months after enrollment
  Parent reported measure of family environment; Reverse odd questions, Average of all question: 1>x<4; Higher scores indicate more problematic perception of family function.
Patient-Reported Outcomes Information System- Short Forms (PROMIS) | At enrollment and approximately 3 months after enrollment
  A bank of measures that examine aspects of individuals' physical, social, and mental health; Average of questions 1>x<5 (Higher scores indicated more perceived support)
FoH-C Frequency of Help | At enrollment and approximately 3 months after enrollment
  10 item assessment of who provides support in the home for diabetes management tasks; Average of items: 1>x>5; higher scores indicate greater frequency of help

CONTACTS AND LOCATIONS:
Locations (1):
- University of California-Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hughes Lansing A, Cohen LB, Glaser NS, Loomba LA. Feasibility and Acceptability of a Self-Guided Digital Family Skills Management Intervention for Children Newly Diagnosed With Type 1 Diabetes: Pilot Randomized Controlled Trial. JMIR Form Res. 2024 Oct 21;8:e59246. doi: 10.2196/59246. PMID 39432892